CLINICAL TRIAL: NCT03238508
Title: Index of Microcirculatory Resistance After Immediate Versus Deferred Stenting in Patients With Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sejong General Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jong Lee, Principle Investigator, Sejong General Hospital
Other Study IDs: Sejong_IRB_1732
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Acute Myocardial Infarction
Keywords: Deferred stenting; Microvascular dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate stenting group: Conventional stenting immediate after the re-opening of infarct-related artery during primary PCI
- Deferred stenting group: Elective stenting following cooling down of infarct- related artery for several days after restoration of epicardial coronary blood flow during primary PCI
  Interventions: Procedure: Deferred stenting

INTERVENTIONS:
Procedure: Deferred stenting — Previously described
  Groups: Deferred stenting group

SUMMARY:
This study will compare the microcirculatory resistance (IMR) of infarct-related artery (IRA) in patients who underwent immediate versus deferred stenting during percutaneous coronary intervention (PCI) for acute myocardial infarction.

DETAILED DESCRIPTION:
Primary PCI with immediate stenting (IS) is the current standard of reperfusion strategy for STEMI. However, it is thought that IS may cause additional myocardial injury by increasing distal embolization of clot and atheromatous plaque debris. Only about 35% of patients without cardiogenic shock can achieve optimal myocardial tissue perfusion at the microvascular level, even after restoration of epicardial coronary artery patency. IS in highly pro-thrombotic and inflammatory milieu of IRA during primary PCI would increase distal embolization of clot and atheromatous plaque debris, and provoke the inflammation process, so deferred stenting after a cooling down period of IRA for several days, have a potential to mitigate or prevent microvascular obstruction (MVO). Among several methods to evaluate MVO after STEMI, IMR has been well known as an good indicator of MVO and strong predictor for short and long term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. More than 30 minutes in duration of typical chest pain
2. Thrombolysis In Myocardial Infarction (TIMI) flow 0, 1 or 2 prior to the procedure

Exclusion Criteria:

1. Cardiogenic shock,
2. Previous history of myocardial infarction, or coronary artery bypass surgery
3. Rescue PCI after fibrinolysis
4. Life expectancy of less than 1 year
5. Acute occlusion of left main coronary artery
6. STEMI due to stent thrombosis
7. Major coronary dissection (type D~F) following procedures achieving TIMI 3 flow

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary precutaneous coronary intervention for ST- segment elevation or Non ST-segment elevation myocardial infarcation with ongoing myocardial ischemia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-08-30 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Index of microcirculatory resistance of infarct-related artery | 3 to 5 days after primary reperfusion (TIMI 3 flow achievement) in both groups
  Measured by pressure and temperature sensors- tipped guide wire

SECONDARY OUTCOMES:
The rate of urgent revascularization | During index hospitalization (intraoperative)
Major bleeding | During index hospitalization (intraoperative)
  Defined as TIMI bleeding criteria
Major adverse cardiac events | One- year after primary reperfusion
  Death, myocardial infarction, unplanned target vessel revascularization or CHF admission

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jong Lee, MD, Principal Investigator — Sejong General Hospital
Locations (1):
- Sejong general hospital, 91-121 Sosa 2-Dong, Sosa-Gu, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JS, Lee HJ, Woong Yu C, Kim YM, Hong SJ, Park JH, Choi RK, Choi YJ, Park JS, Kim TH, Jang HJ, Joo HJ, Cho SA, Ro YM, Lim DS. INNOVATION Study (Impact of Immediate Stent Implantation Versus Deferred Stent Implantation on Infarct Size and Microvascular Perfusion in Patients With ST-Segment-Elevation Myocardial Infarction). Circ Cardiovasc Interv. 2016 Dec;9(12):e004101. doi: 10.1161/CIRCINTERVENTIONS.116.004101. PMID 27965296